CLINICAL TRIAL: NCT02889432
Title: Effects of Oral Melatonin on Neurosensory Recovery Following Facial Osteotomies - A Randomised, Controlled Clinical Trial
Brief Title: Effects of Oral Melatonin on Neurosensory Recovery Following Facial Osteotomies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 16-095
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Dentofacial Deformities
MeSH Terms: conditions — Dentofacial Deformities | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Experimental): Oral Melatonin 10mg Taken 30 minutes before bedtime for 3 weeks First dose starts the night before surgery
  Interventions: Drug: Oral Melatonin 10mg
- Placebo (Placebo Comparator): Placebo tabs Taken 30 minutes before bedtime for 3 weeks First dose starts the night before surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Melatonin 10mg
  Arms: Melatonin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Orthognathic surgery is commonly performed for the treatment of dentofacial deformities. Yet, one of the most prevalent and long-term complication encountered is neurosensory disturbance thus impairing sensation to parts of the face. In Hong Kong, it has been reported that in patients receiving orthognathic surgery, 5.9% experience long-term neurosensory disturbance post-surgery.

Melatonin is a neurohormone that is produced and secreted by the pineal gland in the brain. Its main physiological role in humans is to regulate sleep. Oral Melatonin supplements is also used in the management of jetlag and other sleep disorders. Recently, animal and human studies have shown Melatonin to improve tolerance to pain and to have a neuroprotective and neuroregenerative effect after nerve injuries.

Hence, it is hypothesized that peri-surgical oral Melatonin supplement can improve neurosensory recovery after orthognathic surgery

DETAILED DESCRIPTION:
Background:

Orthognathic surgery is a commonly accepted treatment modality for the management of dentofacial deformities. Although in many cases, satisfying, if not excellent, aesthetic and functional results can be obtained with orthognathic surgeries, this is not without risks; and one of the most prevalent and long-term complication encountered is neurosensory disturbance either in the inferior alveolar nerve or the infraorbital nerve depending on the jaw receiving the osteotomy. A systematic review by Jędrzejewski et al. in 2015 reported cranial nerve injury/sensitivity alteration to be the most common complication after orthognathic surgery and is seen in 50% of cases, and almost all patients will report altered sensation in the immediate post-operative period. Although this will decrease over time, Henzelka et al. have reported a 3% incidence of paresthesia in the inferior alveolar nerve 1 year post-surgery, and Thygesen et al. reported sensory changes in the infraorbital nerve in 7 to 60% of patients depending on site of measurement 1 year post-surgery. In Hong Kong, a 10-year retrospective study of 581 patients by Lee et al. in 2013 reported a 5.9% rate of neurosensory disturbance 1-year post-orthognathic surgery. Of these cases, the majority affected the inferior alveolar nerve, and the combination of ramus osteotomies together with anterior mandibular osteotomies significantly increased the chances of permanent neurosensory disturbance.

Biosynthesis of Melatonin:

Melatonin (N-acetyl-5-methoxytryptamine) is a neurohormone that is endogenously produced and secreted by the pineal gland in the brain in a circadian rhythm, with a plasma concentration highest at night and lowest during the day. Its normal physiological roles in humans are to regulate diurnal rhythm, sleep, mood, immunity, reproduction, intestinal motility, and metabolism. Oral exogenous melatonin has been used in the management of jetlag and other sleep disorders. Recently, animal and human studies have shown melatonin to improve tolerance to tourniquet pain in patients receiving hand surgery performed under regional anaesthesia, to improve dyspnea in patients with chronic obstructive pulmonary disease, and to have a neuroprotective and neuroregenerative effect after nerve injuries.

Pharmacology of Melatonin:

i) Bioavailability: The absorption and bioavailability after oral intake of Melatonin varies greatly. Absorption of Melatonin can range from complete in younger patients and decrease to approximately 50% in the elderly. Bioavailability is usually approximately 15% due to variations in first-pass metabolism. Peak value is ususally observed 60 - 150min after oral consumption. When applied topically to the skin, it has been found that topical application of 0.01% Melatonin cream will increase serum levels of Melatonin from a mean of 4.9pg/mL pre-application to 5.1pg/mL 1-hour post-application to 8.1pg/mL 8-hours post-application, and to 9.0pg/mL 24-hours post-application.

ii) Distribution: Melatonin is highly lipid-soluble with a protein binding capacity of approximately 60%. In vitro, Melatonin has been shown to mainly bind to albumin, alpha1-acid glycoprotein and high-density lipoprotein. Due to its high lipid-solubility, Melatonin has the ability to cross most membrane barriers, including the blood-brain barrier and placenta and can be found in saliva, serum, and urine after oral administration. Melatonin receptors can be found in many tissues throughout the body.

iii) Biotransformation and Excretion: Melatonin is mainly hydroxylated by cytochrome P450 (CYP1A2) in the liver into 6-hydroxymelatonin with a small amount into the serotonin metabolites cyclic 3-hydroxymelatonin and indolinone tautomer of 2-hydroxymelatonin. These are further conjugated to their sulfate and glucuronide conjuates and excreted in the urine.

Usages of Melatonin:

Aside from the regulating sleep and diurnal rhythm, exogenous Melatonin has been recently proved in animal studies and randomized controlled trials in humans to be beneficial in many other areas of medicine and surgery, mostly hypothesized to be due to its antioxidative properties that reduce inflammatory mediators.

A randomized controlled trial by Mowafi and Ismail in 2008 have shown that in patients who required hand surgery with the use of tourniquet under regional anaesthesia, pre-medication with 10mg oral Melatonin 90 minutes before surgery can significanly reduce verbal pain score for tourniquet pain when compared to the placebo group. The time to the first dose of post-operative analgesic request was significantly longer in the Melatonin group and the amount of post-operative analgesic consumption in the Melatonin group was also significantly lower. No significant difference in the incidence of adverse effects between the Melatonin and placebo groups was reported in the study.

Animal studies have shown neuroregenerative and neuroprotective effects of Melatonin. In a controlled study in rats, Atik et al. have shown Melatonin to be beneficial in promoting nerve recovery at high doses. In this study, the tibial and peroneal branches of the sciatic nerve were dissected and subsequently coapted with prolene suture. Post-trauma, 10mg/kg Melatonin was injected intraperitoneally for 21 days. Histologically, rats which received Melatonin exhibited less endoneural collagen with better organizad collagen along the repair line of the nerve. There were also fewer demyelinized axons. By 12 weeks post-trauma, walking track analysis showed significantly better function in the Melatonin group when measured with the sciatic function index (SFI). Electrophysiological findings showed that by 12 weeks post-trauma, the latency was significantly less in the Melatonin group, whilst action potential amplitude and nerve conduction velocity were significantly higher in the Melatonin group compared to the control group. It was concluded in this study that high doses of Melatonin has a significant beneficial effect on nerve recovery as measured functionally, histopathologically, and electrophysiologically.

In another controlled study in rats, Kaya et al. have shown beneficial effects of Melatonin on cut and crush injured sciatic nerve. In this study Melatonin was administered intraperitoneally at a dose of 50mg/kg/day for 6 weeks post-trauma. In terms of SFI values, Melatonin treatment accelerated the recovery process to reach -50 SFI level by the 3rd week, as compared to the placebo group, which only reached this SFI level by the 6th week. Histologically, rats treated with Melatonin showed better strutural preservation of the myelin sheaths compared to the control group. Biochemically, the beneficial effects of Melatonin was further comfirmed by showing lower lipid peroxidation and higher superoxide dismutase, catalase, and glutathione peroxidase activities in sciatic nerve samples when compared to the control group.

Similar beneficial effects were reported by Zencirci et al. in their study of Melatonin in peripheral nerve crush injury in rats. In their study, rats were allocated into the control group or into the treatment group, which further divided into a group receiving 5mg/kg intraperitoneal Melatonin for 21 days post-trauma, and another group receiving 20mg/kg for the same length of time. Again, they have shown an increase in SFI values in the injured sciatic nerves treated with Melatonin when compared to the control group. Electrophysiological measurements again showed that Melatonin treatment deceased the latency values and increased the conduction velocities. However, it was not mentioned whether significant differences were observed between the group receiving 5mg/kg Melatonin and 20mg/kg Melatonin.

Fujimoto et al. were also able to show a potent protective effect of Melatonin on spinal cord injury. In this study, experimental ischemic-induced spinal cord injury was inflicted in rats. Subesequently, the rats were either placed in the controlled group or received 2.5mg/kg Melatonin injected intraperitoneally at 5 minutes, then 1, 2, 3, and 4 hours after injury. It was found that Melatonin reduced the occurrence of neutrophil-induced lipid peroxidation. Melatonin also reduced thiobarbituric acid reactive substance content and myeloperoxidase activity, which were responsible for motor deficits. Histologically, findings from the Melatonin group showed less cavity formation than the control group.

ELIGIBILITY:
Inclusion Criteria:

* No systemic neuropathies
* Clear medical history
* Patients requiring bilateral sagittal split osteotomies, Hofer osteotomy, genioplasty, and/or Le-Fort I osteotomies

Exclusion Criteria:

* Patients with existing neurosensory deficit at the inferior alveolar nerve and/or infraorbital nerve from previous trauma or systemic condition
* Patients with iatrogenic severance of nerve intra-operatively
* Patients who underwent previous orthognathic surgery (i.e. reoperation)
* Patients undergoing distraction osteogenesis
* Patients who developed allergic reactions

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Subjective neurosensory disturbance | Baseline
  VAS score of numbness / hyperaesthesia
Subjective neurosensory disturbance | Post-operative 1 week
  VAS score of numbness / hyperaesthesia
Subjective neurosensory disturbance | Post-operative 1 month
  VAS score of numbness / hyperaesthesia
Subjective neurosensory disturbance | Post-operative 3 months
  VAS score of numbness / hyperaesthesia
Subjective neurosensory disturbance | Post-operative 6 months
  VAS score of numbness / hyperaesthesia
Objective neurosensory disturbance | Baseline
  Static light touch with Von Frey fibres; two-point discrimination; pin-prick pressure
Objective neurosensory disturbance | Post-operative 1 week
  Static light touch with Von Frey fibres; two-point discrimination; pin-prick pressure
Objective neurosensory disturbance | Post-operative 1 month
  Static light touch with Von Frey fibres; two-point discrimination; pin-prick pressure
Objective neurosensory disturbance | Post-operative 3 months
  Static light touch with Von Frey fibres; two-point discrimination; pin-prick pressure
Objective neurosensory disturbance | Post-operative 6 months
  Static light touch with Von Frey fibres; two-point discrimination; pin-prick pressure
Biochemical analysis | Baseline
  Concentration of lipid peroxidase, superoxide dismutase, catalase, and glutathione peroxidase in plasma
Biochemical analysis | Post-operative day 2
  Concentration of lipid peroxidase, superoxide dismutase, catalase, and glutathione peroxidase in plasma

SECONDARY OUTCOMES:
Pain | Post-operative day 0
  VAS pain score; time to first analgesic intake and dosage
Pain | Post-operative day 1
  VAS pain score
Pain | Post-operative day 2
  VAS pain score
Pain | Post-operative day 3
  VAS pain score

CONTACTS AND LOCATIONS:
Overall Officials: Crystal TY Lee, BDS (HKU), Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jedrzejewski M, Smektala T, Sporniak-Tutak K, Olszewski R. Preoperative, intraoperative, and postoperative complications in orthognathic surgery: a systematic review. Clin Oral Investig. 2015 Jun;19(5):969-77. doi: 10.1007/s00784-015-1452-1. Epub 2015 Mar 26. PMID 25804886
- [Background] Mowafi HA, Ismail SA. Melatonin improves tourniquet tolerance and enhances postoperative analgesia in patients receiving intravenous regional anesthesia. Anesth Analg. 2008 Oct;107(4):1422-6. doi: 10.1213/ane.0b013e318181f689. PMID 18806063
- [Background] Atik B, Erkutlu I, Tercan M, Buyukhatipoglu H, Bekerecioglu M, Pence S. The effects of exogenous melatonin on peripheral nerve regeneration and collagen formation in rats. J Surg Res. 2011 Apr;166(2):330-6. doi: 10.1016/j.jss.2009.06.002. Epub 2009 Jul 10. PMID 20006352
- [Background] Kaya Y, Sarikcioglu L, Aslan M, Kencebay C, Demir N, Derin N, Angelov DN, Yildirim FB. Comparison of the beneficial effect of melatonin on recovery after cut and crush sciatic nerve injury: a combined study using functional, electrophysiological, biochemical, and electron microscopic analyses. Childs Nerv Syst. 2013 Mar;29(3):389-401. doi: 10.1007/s00381-012-1936-0. Epub 2012 Oct 9. PMID 23053363
- [Background] Zencirci SG, Bilgin MD, Yaraneri H. Electrophysiological and theoretical analysis of melatonin in peripheral nerve crush injury. J Neurosci Methods. 2010 Aug 30;191(2):277-82. doi: 10.1016/j.jneumeth.2010.07.008. Epub 2010 Jul 14. PMID 20637233
- [Background] Fujimoto T, Nakamura T, Ikeda T, Takagi K. Potent protective effects of melatonin on experimental spinal cord injury. Spine (Phila Pa 1976). 2000 Apr 1;25(7):769-75. doi: 10.1097/00007632-200004010-00003. PMID 10751286
- [Background] de Matos Cavalcante AG, de Bruin PF, de Bruin VM, Nunes DM, Pereira ED, Cavalcante MM, Andrade GM. Melatonin reduces lung oxidative stress in patients with chronic obstructive pulmonary disease: a randomized, double-blind, placebo-controlled study. J Pineal Res. 2012 Oct;53(3):238-44. doi: 10.1111/j.1600-079X.2012.00992.x. Epub 2012 Apr 17. PMID 22507631
- [Background] Odaci E, Kaplan S. Chapter 16: Melatonin and nerve regeneration. Int Rev Neurobiol. 2009;87:317-35. doi: 10.1016/S0074-7742(09)87016-5. PMID 19682645
- [Background] Kleszczynski K, Fischer TW. Melatonin and human skin aging. Dermatoendocrinol. 2012 Jul 1;4(3):245-52. doi: 10.4161/derm.22344. PMID 23467217
- [Background] Di WL, Kadva A, Johnston A, Silman R. Variable bioavailability of oral melatonin. N Engl J Med. 1997 Apr 3;336(14):1028-9. doi: 10.1056/NEJM199704033361418. No abstract available. PMID 9091795
- [Background] Waldhauser F, Waldhauser M, Lieberman HR, Deng MH, Lynch HJ, Wurtman RJ. Bioavailability of oral melatonin in humans. Neuroendocrinology. 1984 Oct;39(4):307-13. doi: 10.1159/000123997. PMID 6493445
- [Background] Fischer TW, Greif C, Fluhr JW, Wigger-Alberti W, Elsner P. Percutaneous penetration of topically applied melatonin in a cream and an alcoholic solution. Skin Pharmacol Physiol. 2004 Jul-Aug;17(4):190-4. doi: 10.1159/000078822. PMID 15258450
- [Background] Vakkuri O, Leppaluoto J, Kauppila A. Oral administration and distribution of melatonin in human serum, saliva and urine. Life Sci. 1985 Aug 5;37(5):489-95. doi: 10.1016/0024-3205(85)90412-6. PMID 4021725
- [Background] Ma X, Idle JR, Krausz KW, Gonzalez FJ. Metabolism of melatonin by human cytochromes p450. Drug Metab Dispos. 2005 Apr;33(4):489-94. doi: 10.1124/dmd.104.002410. Epub 2004 Dec 22. PMID 15616152